CLINICAL TRIAL: NCT05214274
Title: The Status of Diagnosis and Treatment of Chronic Hypoparathyroidism in Chinese Adults: a Multicenter Registry Study
Brief Title: Multicenter Registry Study of Chronic Hypoparathyroidism in Chinese Adults
Acronym: PaTHwayR
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Collaborators: Peking Union Medical College Hospital (Other); Shanghai 6th People's Hospital (Other); First Hospital of China Medical University (Other); Central South University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); West China Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-PaTHwayR
Record Dates: First submitted 2021-12-24; First posted 2022-01-28 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Chronic Hypoparathyroidism
Keywords: Registry study; Chronic hypoparathyroidism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention would be taken — No intervention would be taken

SUMMARY:
This multicenter registry study aims to understand the status of diagnosis and treatment, quality of life, medical costs and unmet medical needs of adult patients with chronic hypoparathyroidism in China.

DETAILED DESCRIPTION:
Hypoparathyroidism (HP) is a rare (orphan) endocrine disease with low calcium and inappropriately low circulating parathyroid hormone levels, most often in adults secondary to thyroid surgery. The present study contains four parts.

The first part is a multicenter registry study. According to our predefined search criteria determined through pilot study, all patients admitted between June 1, 2020 and May 31, 2021 will be searched from the hospital information system and patients diagnosed with HP and those with suspected HP will be retrieved. The diagnosis of all or a random sample of these patients will be reviewed by endocrinologists through medical records. Patients with a confirmed diagnosis of chronic HP will served as the study population of the first part of the study.

The second part is a multicenter hospital-based survey, to investigate the missed diagnosis, quality of life, medical costs, medical experience and unmet medical needs in adult patients with chronic HP. All local patients with definite chronic HP and those with suspected HP will be invited to participate in the hospital on-site investigation. Among them, suspected HP patients need to first undergo necessary examinations to confirm the diagnosis of HP.

The third part is the verification of the reliability and validity of two quality of life scales, the Short-Form Six-Dimension version 2 (SF-6Dv2) scale and Hypoparathyroidism Patient Experience Scale (HPES). The first 100 patients with chronic HP who participate in the on-site investigation in the Peking Union Medical College Hospital will be invited.

The fourth part is a survey on physicians about the unmet need of chronic HP. All endocrinologists from each site will be invited to take part in the survey.

ELIGIBILITY:
This study consists of four parts, the eligibility criteria of each part is described below:

Part 1:

Search criteria of chronic HP:

Inclusion Criteria:

* Existing diagnosis of HP

Exclusion Criteria:

* Age<18 at the time of screening

Search criteria of suspected HP:

Inclusion Criteria:

* Hypocalcemia plus neck surgery
* Hypocalcemia plus convulsions/tetany/epilepsy
* Hypocalcemia plus PTH<upper limit, and no hypoalbuminemia
* Hypocalcemia without any of the following conditions: neck surgery, convulsions/tetany/epilepsy, PTH testing, hypoalbuminemia, critical illness and vitamin D deficiency-related diseases.

Exclusion Criteria:

* Age<18 at the time of screening

Diagnosis of chronic HP:

Inclusion Criteria:

* Hypocalcemia (albumin adjusted total calcium < lower limit) with inappropriate reduction of serum PTH level (PTH < upper limit).
* The course of hypoparathyroidism should be more than 6 months.

Part 2

Inclusion Criteria:

* Patients with chronic HP confirmed through medical records review
* Patients with suspected HP confirmed through medical records review
* Obtain written informed consent

Exclusion Criteria:

* Non-local residents

Part 3

Inclusion Criteria:

* Patients with chronic HP
* Participating in the on-site survey in the Peking Union Medical College Hospital

Part 4

Inclusion criteria:

* Endocrinologists involved in HP care from 7 sites
* Obtain written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Part 1. All patients admitted between June 1, 2020 and May 31, 2021 will be searched in the information system according to predefined search criteria. Patients diagnosed with HP and those with suspected HP will be retrieved. Patients with definite diagnosis of chronic HP will serve as the study population of this part.
  Part 2. All local patients with a definite diagnosis of chronic HP and those with suspected HP will be invited to take part in the on-site survey.
  Part 3. The first 100 patients with definite chronic HP who participate in the on-site survey in the Peking Union Medical College Hospital will be invited to participate.
  Part 4. All endocrinologists at each center will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with different classification of hypoparathyroidism (HP) | 0 day （cross-sectional）
  HP is classified into postsurgical and non-postsurgical HP.
The proportion of patients with different symptoms of HP | 0 day （cross-sectional）
  The most common symptoms of HP include tetany, seizures, laryngospasm, numbness, blood in the urine, renal colic and vision loss.
The proportion of patients with positive Chvostek sign | 0 day （cross-sectional）
  Including the situation at the time of diagnosis and the current situation
The proportion of patients with positive Trousseau's sign | 0 day （cross-sectional）
  Including the situation at the time of diagnosis and the current situation
The proportion of patients with abnormal corrected calcium | 0 day （cross-sectional）
  Including the situation at the time of diagnosis and the current situation
The proportion of patients with abnormal parathyroid hormone (PTH) | 0 day （cross-sectional）
  The situation at the time of diagnosis
The proportion of patients with abnormal 24-hour urine calcium | 0 day （cross-sectional）
  Including the situation at the time of diagnosis and the current situation
The proportion of patients with different first-visit reasons | 0 day （cross-sectional）
  First-visit reason was excerpted from previous medical records
The proportion of patients with different first-visit departments | 0 day （cross-sectional）
  First-visit department was excerpted from previous medical records

SECONDARY OUTCOMES:
The prevalence of chronic HP in adults visiting top hospitals in China | 0 day （cross-sectional）
  Number of patients diagnosed with chronic HP / Total number of outpatients and inpatients during the year
The proportion of patients with chronic HP receiving treatment | 0 day （cross-sectional）
  Number of patients receiving any kind of HP treatment/ Total number of patients diagnosed with chronic HP
The proportion of patients with chronic HP meeting treatment targets | 0 day （cross-sectional）
  HP treatment targets defined as normal blood calcium levels or/+ normal urine calcium level
The proportion of patients with HP complications | 0 day （cross-sectional）
  Number of patients with complications / Total number of patients with chronic HP
The proportion of patients with missed diagnosis of chronic HP | 0 day （cross-sectional）
  Patients with missed diagnosis of chronic HP / Total number of patients with chronic HP
The proportion of patients with previous experience of misdiagnosis of HP | 0 day （cross-sectional）
  Misdiagnosis experience of HP is defined as patients with chronic HP were previously diagnosed with other diseases due to related symptoms or hypocalcemia.
Median medical costs | 0 day （cross-sectional）
  Medical costs contains of direct medical costs and indirect medical costs
The mean score of Short-Form Six-Dimension version 2 (SF-6Dv2) | 0 day （cross-sectional）
  The SF-6Dv2 score ranges from 0.29 to 1, with higher scores indicating better performance.
The mean score of Hypoparathyroidism Patient Experience Scale (HPES) | 0 day （cross-sectional）
  The HPES score ranges from 0 to 100, with lower scores indicating better performance.
The proportion of patients with different unmet medical needs | 0 day （cross-sectional）
  Unmet medical needs for HP treatment and quality of life by patients and physicians

CONTACTS AND LOCATIONS:
Overall Officials: Weibo Xia, Principal Investigator — Peking Union Medical College Hospital
Locations (7):
- China (7):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Hospital of China Medical University, Shenyang, Dongbei
  - The First Affiliated Hospital , Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: Undecided